CLINICAL TRIAL: NCT01349673
Title: A Phase 3, Open Label, Multicenter Study to Assess the Safety and Tolerability of Budesonide Foam in Subjects With Active Ulcerative Proctitis or Proctosigmoiditis
Brief Title: The Safety and Tolerability of Budesonide Foam in Participants With Active Ulcerative Proctitis or Proctosigmoiditis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated for non-safety reasons when Sponsor felt that sufficient long-term safety data was obtained.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFPS3073
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Proctitis; Proctosigmoiditis
Keywords: Open-label; Proctitis; Proctosigmoiditis; Ulcerative; Salix; Budesonide foam; Budesonide; Rectal; Gastrointestinal; Colitis; UC; UP; UPS; Additional relevant MeSH terms:; Proctocolitis; Ulcer; Colitis, Ulcerative; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Rectal Diseases; Intestinal Diseases; Colonic Diseases; Sigmoid Diseases; Pathologic Processes; Inflammatory Bowel Diseases; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Physiological Effects of Drugs; Pharmacologic Actions; Anti-Asthmatic Agents; Respiratory System Agents; Therapeutic Uses; Glucocorticoids; Hormones; Hormones, Hormone Substitutes and Hormone Antagonists; Anti-inflammatory Agents
MeSH Terms: conditions — Proctitis; Proctocolitis; Ulcer; Colitis; Colitis, Ulcerative; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Rectal Diseases; Intestinal Diseases; Colonic Diseases; Sigmoid Diseases; Pathologic Processes; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Budesonide Foam (Experimental): Participants administered topical rectal budesonide foam at 2 mg/25 mL BID (morning and 12 hours later) for 2 weeks followed by 2 mg/25 mL QD (in the evenings) for 4 weeks for up to 8 cycles. After Cycle 1, participants needed to qualify to be able to participate in subsequent cycles. Participants underwent a 48-hour study drug washout period between each cycle.
  Interventions: Drug: Budesonide Foam

INTERVENTIONS:
Drug: Budesonide Foam — Topical

SUMMARY:
The purpose of this study is to evaluate safety and tolerability of cyclically-dosed rectal budesonide foam in participants with active ulcerative proctitis (UP) or ulcerative proctosigmoiditis (UPS).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, open-label study in participants who previously participated in a Salix-sponsored budesonide rectal foam study for the treatment of UP or UPS. Approximately 300 participants were to be enrolled into the study and receive budesonide foam cyclically for 6 weeks (twice a day [BID] for 2 weeks and once daily [QD] for 4 weeks). The study was to continue until regulatory approval of budesonide foam occurred or the sponsor decided to terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-breast-feeding females ≥18 years old.
* Participant was previously diagnosed with active mild to moderate UP/UPS and was currently experiencing symptoms of active UP/UPS disease after having completed participation in Salix's BUCF3001 (NCT01008410) or BUCF3002 (NCT01008423) study.
* Willingness to undergo sigmoidoscopy.

Exclusion Criteria:

* Active systemic, ocular, or cutaneous infection (for example, parasitic, fungal, amoebic, viral, or bacterial disease).
* History of sclerosing cholangitis, cirrhosis, or hepatic impairment, including chronic hepatitis of any etiology.
* Participant took systemic, inhaled, oral, topical, or rectal corticosteroids (other than budesonide rectal foam) within 7 days of starting a treatment cycle.
* Participant took ketoconazole and other potent CYP3A4 inhibitors within 7 days of starting a treatment cycle.
* Participant took diuretics with cardiac glycosides.
* Unstable significant cardiovascular, hepatic, renal, endocrine, neurologic, or pulmonary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Consultants, PA, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant received study drug for 6 weeks per cycle for up to 8 cycles and underwent a 48-hour study drug washout period between each cycle. Study was terminated for non-safety reasons when Sponsor felt sufficient long-term safety data was obtained.
Period: Overall Study
Arm/Group | Budesonide Foam
Started | 114
Participants Entered Cycle 1 | 114
Participants Entered Cycle 2 | 65
Participants Entered Cycle 3 | 41
Participants Entered Cycle 4 | 22
Participants Entered Cycle 5 | 12
Participants Entered Cycle 6 | 5
Participants Entered Cycle 7 | 3
Participants Entered Cycle 8 | 1
Received At Least 1 Dose Of Study Drug | 114
Completed | 0
Not Completed | 114
Not completed — Progression Of Disease Past 40 cm | 1
Not completed — No Longer Qualified For Study | 1
Not completed — Site Closure | 10
Not completed — Withdrawal by Subject | 21
Not completed — Lost to Follow-up | 6
Not completed — Adverse Event | 17
Not completed — Study Terminated By Sponsor | 50
Not completed — Lack of Efficacy | 8

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Arm/Group | Budesonide Foam
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Reporting A Non-serious Adverse Event And A Serious Adverse Event
Description: A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through up to Cycle 8 (Cycle=6 weeks)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide Foam
Number analyzed (Participants) | 114
Participants
  Non-serious Adverse Event | 66
  Serious Adverse Event | 0

2. Secondary Outcome: Clinically Notable Laboratory Parameters
Description: Clinically notable laboratory parameters are defined as clinical laboratory values outside the reference range. Reference ranges for the clinical notable laboratory parameters: Aspartate Aminotransferase - 0-37 microliters (U/L); Alanine Aminotransferase - 0-47 U/L; Lactate Dehydrogenase - 110-250 U/L. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline and Cycle 4 (Cycle=6 weeks)
Population: All participants who received at least 1 dose of study drug and with non-missing clinical laboratory parameter values at the specified timepoint.
Measure: Mean (Full Range); unit: U/L
Arm/Group | Budesonide Foam
Number analyzed (Participants) | 114
U/L
  Aspartate Aminotransferase, Baseline | 21.7 [12 to 37]
  Aspartate Aminotransferase, Cycle 4: number analyzed (Participants) | 6
  Aspartate Aminotransferase, Cycle 4 | 92.3 [21 to 440]
  Alanine Aminotransferase, Baseline | 23.0 [7 to 58]
  Alanine Aminotransferase, Cycle 4: number analyzed (Participants) | 6
  Alanine Aminotransferase, Cycle 4 | 119.3 [13 to 596]
  Lactate Dehydrogenase, Baseline | 154.1 [82 to 223]
  Lactate Dehydrogenase, Cycle 4: number analyzed (Participants) | 6
  Lactate Dehydrogenase, Cycle 4 | 228.5 [143 to 506]

3. Secondary Outcome: Changes In Baseline In Mean Morning (AM) Fasting Serum Cortisol Levels
Description: Fasting cortisol levels were evaluated, and cortisol was taken in the morning (AM cortisol) approximately 2 to 4 hours after waking. Data for cycles with more than 15 participants at the Cycle Baseline is reported.
Time Frame: Baseline of Cycles 1-4, Day 15 and Day 42 of Cycles 1-4 (Cycle=6 weeks)
Population: All participants who received at least 1 dose of study drug and with non-missing cortisol value at the specified timepoint.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Budesonide Foam
Number analyzed (Participants) | 114
nanomoles per liter (nmol/L)
  Cycle 1, Day 15: number analyzed (Participants) | 104
  Cycle 1, Day 15 | -62.7 (149.61)
  Cycle 1, Day 42: number analyzed (Participants) | 90
  Cycle 1, Day 42 | 0.9 (170.78)
  Cycle 2, Day 15: number analyzed (Participants) | 60
  Cycle 2, Day 15 | -40.1 (165.65)
  Cycle 2, Day 42: number analyzed (Participants) | 52
  Cycle 2, Day 42 | -5.8 (183.16)
  Cycle 3, Day 15: number analyzed (Participants) | 34
  Cycle 3, Day 15 | -25.5 (175.75)
  Cycle 3, Day 42: number analyzed (Participants) | 31
  Cycle 3, Day 42 | -10.4 (174.92)
  Cycle 4, Day 15: number analyzed (Participants) | 20
  Cycle 4, Day 15 | -87.8 (186.11)
  Cycle 4, Day 42: number analyzed (Participants) | 16
  Cycle 4, Day 42 | -7.1 (148.52)

4. Secondary Outcome: Number of Participants With A Clinically Notable Physical Examination Finding Since Baseline
Description: A full or complete physical examination was performed at the Study Baseline. This physical examination included (but was not limited to): general appearance, head, ear, eyes, nose, throat, respiratory, cardiovascular, gastrointestinal, abdominal, neurological, lymphatic, dermatologic, and musculoskeletal. A symptom-directed physical examination was performed on Visit 2 (Day 1) to Visit 4 (Day 42) per Cycle (at the Investigator's discretion) and as needed for unscheduled clinic visits. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through up to Cycle 8 (Cycle=6 weeks)
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Budesonide Foam
Number analyzed (Participants) | 114
Participants | 17

ADVERSE EVENTS:
Time Frame: Baseline through up to Cycle 8 (Cycle=6 weeks)
Arm/Group | Budesonide Foam
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 66/114
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide Foam (N=114)
Adrenal insufficiency (Endocrine disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 9
Anorectal discomfort (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Colitis ulcerative (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Nasopharyngitis (Infections and infestations) | 4
Blood cortisol decreased (Investigations) | 20
Headache (Nervous system disorders) | 8
Depression (Psychiatric disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.